CLINICAL TRIAL: NCT05095623
Title: A Natural History Study to Assess the Clinical Outcomes of Patients With Complement Factor I Deficiency-Mediated Disease
Status: Terminated | Type: Observational
Why Stopped: enrollment
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: CFI-002
Record Dates: First submitted 2021-09-29; First posted 2021-10-27 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Bacterial Infection, Autoimmune Disorder
MeSH Terms: conditions — Bacterial Infections; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Natural History Observation — This is a natural history study.

SUMMARY:
This study will follow participants with a disease which is associated with an absence or deficiency in Complement Factor I (CFI) as confirmed in the CFI-001 screening study.

DETAILED DESCRIPTION:
This study will follow participants with a disease which is associated with an absence or deficiency in Complement Factor I (CFI) as confirmed in the CFI-001 screening study.

The population will include male and female participants ≥6 months of age (pediatric participants enrolled as permitted by local Institutional Review Board/Independent Ethics Committee). This includes patients with recurrent bacterial infections (eg, meningitis, sepsis, pneumonia, endocarditis, otitis) and patients with autoimmune and immune complex-mediated diseases (eg, glomerulonephritis, systemic lupus erythematosus, leukocytoclastic vasculitis, Bickerstaff encephalitis, meningoencephalitis).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 6 months or older
2. Affirmation of participant's informed consent or legally authorized representative (LAR)'s willingness to provide informed consent with signature confirmation before any study-related activities. (Study-related activities are any procedures that would not have been performed during normal clinical management of the participant.) The participant (if a minor) must also be willing to give written informed assent (if able) if the minor is within the age groups 7 to 11 years old and 12 to 17 years old.
3. Confirmed CFI deficiency during the screening study, CFI-001, with a disease that is associated with an absence or deficiency in CFI
4. Stated willingness of the participant to comply with all study procedures (including multiple blood draws) and availability for the duration of the study
5. Stated willingness of the participant (or LAR) to allow access to his/her medical records with the purpose of assessing disease status and progression during his/her participation in the study

Exclusion Criteria:

1. Participation in an interventional clinical study within the previous 30 days prior to screening or within ≤5 half-lives of the investigational drug, whichever is longer
2. Having a major concurrent non-CFI-related disease that prevents the assessment of the natural course of the CFI deficiency disease
3. Having a medical, psychosocial, or familial issues that might prevent full participation and cooperation with the procedures and requirements of the clinical study as determined by the potential participant/guardian and physician investigator

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will follow participants with a disease which is associated with an absence or deficiency in Complement Factor I (CFI) as confirmed in the CFI-001 screening study. The population will include male and female participants ≥6 months of age (pediatric participants enrolled as permitted by local Institutional Review Board/Independent Ethics Committee). This includes patients with recurrent bacterial infections (eg, meningitis, sepsis, pneumonia, endocarditis, otitis) and patients with autoimmune and immune complex-mediated diseases (eg, glomerulonephritis, systemic lupus erythematosus, leukocytoclastic vasculitis, Bickerstaff encephalitis, meningoencephalitis).
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
General clinical condition | Approximately every 3 months
  General clinical condition
Proportion of patients with episodes or exacerbations of medical events | Approximately every 3 months
  Proportion of patients with episodes or exacerbations of medical events
Proportion of patients with infections As applicable, infections (particularly meningococcal and other encapsulated bacteria) | Approximately every 3 months
  Proportion of patients with infections
Proportion of patients with kidney disease progression | Approximately every 3 months
  Proportion of patients with kidney disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Consultants, LLC, Huntsville, Alabama, United States